CLINICAL TRIAL: NCT06679478
Title: Evaluation of the Early Mobilization Protocol Established in Accordance With Enhanced Recovery After Surgery Guidelines in Patients Undergoing Gastrointestinal Surgery
Brief Title: Evaluation of Early Mobilization Protocol in Patients Undergoing Gastrointestinal Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Derya Şayır Koksal, lecturer, Uludag University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UludagU-SBF-DSK-01
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Gastrointestinal Diseases
Keywords: Gastrointestinal Diseases; Enhanced Recovery After Surgery; Early Ambulation
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: The participants in the control group are given the mobilization applied in routine clinics. The participants in the intervention group are given the mobilization protocol created in accordance with the enhanced recovery after surgery guidelines.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants are not informed of which group they are in. The investigators will not inform the person performing the statistical analysis which group the collected data belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization Performed in Routine Clinic Group (No Intervention): Participants undergoing gastrointestinal surgery will receive routine clinic mobilization. The investigator will not perform any interventions.
- Early Mobilization Protocol Created in Enhanced Recovery After Surgery (ERAS) Guidelines Group (Experimental): Participants undergoing gastrointestinal surgery will watch a video 1 day before surgery that includes information about the importance of mobilization and the process.
  The participant will be applied a mobilization protocol created in line with the postoperative mobilization eras (enhanced recovery after surgery) guidelines.
  Interventions: Procedure: Enhanced Recovery After Surgery (ERAS) Early Mobilization Protocol

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery (ERAS) Early Mobilization Protocol — The intervention is applied from the first day after surgery until discharge. (including the day of discharge).
  Other Names: Early Mobilization Protocol
  Arms: Early Mobilization Protocol Created in Enhanced Recovery After Surgery (ERAS) Guidelines Group

SUMMARY:
In this study, the investigators aimed to evaluate the early mobilization protocol created in accordance with the accelerated recovery guide after surgery in patients undergoing gastrointestinal surgery.

DETAILED DESCRIPTION:
This study is an experimental study. The participants in the control group are applied to the mobilization applied in routine clinics. The participants in the intervention group are applied to the mobilization protocol created in accordance with the Enhanced Recovery After Surgery (ERAS) guidelines. It is planned to evaluate the postoperative mobilization process of both groups.

In this study, the researchers aimed to evaluate the early mobilization protocol created in accordance with the accelerated recovery guide after surgery in patients undergoing gastrointestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Agreeing to participate in the study
* Being able to understand, speak Turkish or have no obstacle to communication
* Having undergone open gastrointestinal surgery
* Having an American Society of Anesthesiologists (ASA) score <IV
* Being fully independent according to the Modified Barthel Index during the pre-operative period
* Staying in the hospital for at least 48 hours after the surgery
* Having a phone
* Agreeing to download the 'StepsApp Pedometer' application to their phone
* Agreeing to carry the phone with them during the post-operative mobilization processes

Exclusion Criteria:

* Being taken into emergency surgery
* Having had major gastrointestinal surgery before
* Having a diagnosis that may restrict mobilization (neurological, cardiovascular, respiratory and musculoskeletal comorbidities)
* High risk of falling in the preoperative period
* Using medication that may affect mobilization
* Having a diagnosis of any psychiatric disease
* Having a Nutritional Risk Score score of ≥3
* Being in contact isolation
* Being morbidly obese
* Being in intensive care for more than 24 hours during the postoperative period
* Having an intubation period of more than 24 hours during the postoperative period
* Developing a complication that may prevent mobilization after surgery
* Withdrawing from participating in the study,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-09 (Estimated)

PRIMARY OUTCOMES:
The effect of the ERAS (Enhanced Recovery After Surgery) early mobilization protocol on the number of steps taken daily after surgery | From admission to discharge, up to 1 week
  The number of steps taken by the participant daily after surgery will be measured via a phone pedometer application (StepsApp).
The effect of the ERAS (Enhanced Recovery After Surgery) early mobilization protocol on the distance moved after surgery | From admission to discharge, up to 1 week
  The daily distance moved by the participant after surgery will be measured via a phone pedometer application (StepsApp).
The effect of the ERAS early mobilization protocol on the recovery of the gastrointestinal system after surgery | From admission to discharge, up to 1 week
  The researcher will record the day the participant first passed gas after surgery and the date of his/her first defecation.
The effect of the ERAS (Enhanced Recovery After Surgery) early mobilization protocol on the level of ability to perform daily living activities after surgery | (From admission to discharge, up to 1 week) and (When he comes for a check-up 1 week after discharge)
  The researcher makes the measurement with the Modified Barthel Index scale. Modified Barthel Index: The highest score is 100, the lowest score is 0. The patient is stated as fully dependent in the range of 0-20 points, highly dependent in the range of 21-61 points, moderately dependent in the range of 62-90 points, slightly dependent in the range of 91-99 points, and fully independent in the range of 100 points. Daily evaluations are made until discharge after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Şayır Köksal, Lecturer, Principal Investigator
Locations (1):
- Derya Şayır Köksal, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No